CLINICAL TRIAL: NCT00216203
Title: A Phase I-IIa Dose-Ranging Study of Pemetrexed (Alimta) Plus Cetuximab (Erbitux) in Patients With Recurrent Non-Small Cell Lung Cancer (NSCLC): Hoosier Oncology Group LUN04-79
Brief Title: Pemetrexed Plus Cetuximab in Patients With Recurrent Non Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nasser Hanna, M.D. (Other)
Collaborators: Eli Lilly and Company (Industry); Bristol-Myers Squibb (Industry); Walther Cancer Institute (Other)
Responsible Party: Sponsor-Investigator, Nasser Hanna, M.D., Sponsor-Investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HOG LUN04-79
Record Dates: First submitted 2005-09-12; First posted 2005-09-22 (Estimated); Results first posted 2016-06-02 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-08

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Investigational Treatment (Experimental): Pemetrexed + cetuximab for patients with recurrent non-small cell lung cancer.
  Interventions: Drug: Pemetrexed; Drug: Cetuximab

INTERVENTIONS:
Drug: Pemetrexed — Pemetrexed at the assigned dose, day 1 of each 21 day cycle for a maximum of 6 cycles
Drug: Cetuximab — Cetuximab 400 mg/m2, week 1, day 1
  Cetuximab 250 mg/m2, day 1, 8, 15 of each 21 day cycle

SUMMARY:
Both pemetrexed and cetuximab have single agent activity in NSCLC and non-overlapping toxicity profiles. While 2-drug combination therapy has proven superior to single agent therapy in the first-line setting of NSCLC, no such phase III trials have been reported in the second-line setting. Therefore, the purpose of this study is to determine the feasibility of combining these drugs, assessing the toxicity profile, determining the MTD and evaluating the activity of the combination in an expanded phase II setting. If the combination appears to have promising activity, further evaluation of this regimen may be warranted comparing it to single agent pemetrexed or cetuximab alone.

DETAILED DESCRIPTION:
OUTLINE: This is a multi-center study.

Week 1 (day 1):

* Cetuximab 400mg/m2

Week 2 (Cycle 1, Day 1):

* Cetuximab 250mg/m2 plus premetrexed at the assigned dose level.

Patients will be treated with cetuximab on day 1, 8, 15 of each 21 day cycle.

Patients will be treated with pemetrexed on day 1 of each 21 day cycle for a maximum of 6 cycles.

Acceptable toxicity and SD, PR or CR: treat up to 6 cycles then continue cetuximab weekly until PD or excess toxicity

Performance status: ECOG 0-2

Life expectancy: At least 12 weeks

Hematopoietic:

* ANC > 1,500/mm3
* Platelets > 100,000/mm3

Hepatic:

* Bilirubin less than or equal to the upper limit of normal (ULN)
* Aspartate aminotransferase (AST) < 1.5 X ULN. AST may be < 5 X ULN for patients with liver metastases
* Alkaline phosphatase < 5 X ULN

Renal:

* Calculated creatinine clearance > 45 mL/min (by Cockcroft-Gault)

Cardiovascular:

* No significant history of uncontrolled cardiac disease (i.e., uncontrolled hypertension, unstable angina, and congestive heart failure)

Pulmonary:

* Not specified

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic diagnosis of NSCLC
* Recurrent or metastatic disease that is not amenable to curative therapyMeasurable disease according to RECIST
* At least one prior platinum containing regimen for either locally advanced or metastatic disease
* Prior chemotherapy must be completed at least 21 days prior to being registered for protocol therapy and the subject must have recovered from the acute toxicity effects of the regimen
* Ability and willingness to interrupt aspirin or other nonsteroidal anti-inflammatory agents for a 5-day period
* Prior radiation therapy allowed to < 25% of the bone marrow
* Negative pregnancy test

Exclusion Criteria:

* No active infection that in the opinion of the investigator would compromise the subject's ability to tolerate therapy.
* No serious concomitant systemic disorders that would compromise the safety of the subject or compromise the subject's ability to complete the study, at the discretion of the investigator.
* No prior malignancy is allowed except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the subject has been disease-free for at least 2 years.
* No major thoracic or abdominal surgery within 30 days prior to being registered for protocol therapy.
* No current breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2005-05; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nasser Hanna, M.D., Study Chair — Hoosier Oncology Group, LLC
Locations (11):
- United States (11):
  - Medical & Surgical Specialists, LLC, Galesburg, Illinois
  - Cancer Care Center of Southern Indiana, Bloomington, Indiana
  - Elkhart Clinic, Elkhart, Indiana
  - Fort Wayne Oncology & Hematology, Inc, Fort Wayne, Indiana
  - Center for Cancer Care at Goshen Health System, Goshen, Indiana
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Medical Consultants, P.C., Muncie, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Greenebaum Cancer Center, Baltimore, Maryland
  - Oncology Hematology Care, Inc., Cincinnati, Ohio
  - Texas Oncology Cancer Center, Austin, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jalal S, Waterhouse D, Edelman MJ, Nattam S, Ansari R, Koneru K, Clark R, Richards A, Wu J, Yu M, Bottema B, White A, Hanna N. Pemetrexed plus cetuximab in patients with recurrent non-small cell lung cancer (NSCLC): a phase I/II study from the Hoosier Oncology Group. J Thorac Oncol. 2009 Nov;4(11):1420-4. doi: 10.1097/JTO.0b013e3181b624ae. PMID 19701110
- See also: Hoosier Oncology Group Home Page — http://hoosieroncologygroup.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Pemetrexed + Cetuximab: Pemetrexed + cetuximab for patients with recurrent non-small cell lung cancer.
  Pemetrexed: Pemetrexed at the assigned dose, day 1 of each 21 day cycle for a maximum of 6 cycles
  Cetuximab: Cetuximab 400 mg/m2, week 1, day 1
  Cetuximab 250 mg/m2, day 1, 8, 15 of each 21 day cycle
Period: Overall Study
Arm/Group | Pemetrexed + Cetuximab
Started | 36
Completed | 34
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: 33 of 36 consented participants received treatment.
Arm/Group | Pemetrexed + Cetuximab
Number analyzed (Participants) | 33
Age, Continuous [Median (Full Range); unit: years] | 64 [37 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 20
Region of Enrollment [Number; unit: participants]
  United States | 33
Eastern Cooperative Oncology Group (ECOG) performance status [Number; unit: participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) from 0-5 that describes a patient's level of functioning where 0=Fully active, able to carry on all pre-disease performance without restriction and 5=Dead:
  participants
    ECOG PS 0 | 19
    ECOG PS 1 | 14
Disease Stage [Number; unit: participants] — Stage III: Cancer is present. The higher the number, the larger the cancer tumor and the more it has spread into nearby tissues.
  Stage IV: The cancer has spread to distant parts of the body.
  participants
    Disease Stage III | 2
    Disease Stage IV | 31
Tumor Histology [Number; unit: participants]
  Adenocarcinoma | 18
  Squamous cell carcinoma | 8
  Large cell carcinoma | 2
  Non-small cell carcinoma (NOS) | 5
Smoking History [Number; unit: participants]
  Current Smoker | 6
  Former Smoker | 24
  Never a Smoker | 3
Previous Treatment [Number; unit: participants]
  1 Chemotherapy | 26
  2 Chemotherapy | 5
  >2 Chemotherapy | 2
  Previous Targeted Therapy | 6
  Previous radiotherapy | 14

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Pemetrexed in Combination With Cetuximab
Description: The primary objective of the phase I portion of this study is to define the maximum tolerated dose (MTD) of the combination of pemetrexed and cetuximab
Time Frame: 12 months
Population: 12 participants participated in the phase I portion of the trial.
Measure: Number; unit: mg/m^2 every 21 days
Groups:
- Investigational Treatment: Pemetrexed + cetuximab for patients with recurrent non-small cell lung cancer.
  Pemetrexed: Pemetrexed at the assigned dose, day 1 of each 21 day cycle for a maximum of 6 cycles
  Cetuximab: Cetuximab 400 mg/m2, week 1, day 1
  Cetuximab 250 mg/m2, day 1, 8, 15 of each 21 day cycle
Arm/Group | Investigational Treatment
Number analyzed (Participants) | 12
mg/m^2 every 21 days | 750

2. Primary Outcome: Time To Progression (TTP)
Description: The primary objective of the phase II portion is to estimate the time to progression of this combination, evaluated per RECIST criteria where PD= at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions
Time Frame: 24 Months
Population: 27 participants had enough data to complete TTP analysis
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Pemetrexed + Cetuximab
Number analyzed (Participants) | 27
Weeks | 14.6 [6.0 to 78.7]

3. Secondary Outcome: Median Survival Time
Time Frame: 24 Months
Population: 27 participants had data sufficient to complete Median Survival Time analysis
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Pemetrexed + Cetuximab
Number analyzed (Participants) | 27
weeks | 42.0 [8.6 to 103.9]

4. Secondary Outcome: Toxicity and Safety Profile
Time Frame: 12 months
Measure: Number; unit: percentage of particpants
Arm/Group | Pemetrexed + Cetuximab
Number analyzed (Participants) | 33
percentage of particpants
  Acne-like rash: Phase I - Any Grade | 58.3
  Acne-like rash: Phase I - Grade 3/4 | 16.7
  Acne-like rash: Phase II - Any Grade | 57
  Acne-like rash: Phase II - Grade 3/4 | 23.8
  ALT elevation: Phase I - Any Grade | 33.3
  ALT elevation: Phase I - Grade 3/4 | 16.7
  ALT elevation: Phase II - Any Grade | 0
  ALT elevation: Phase II - Grade 3/4 | 0
  Anemia: Phase I - Any Grade | 0
  Anemia: Phase I - Grade 3/4 | 0
  Anemia: Phase II - Any Grade | 14.3
  Anemia: Phase II - Grade 3/4 | 0
  Thrombocytopenia: Phase I - Any Grade | 8.3
  Thrombocytopenia: Phase I - Grade 3/4 | 0
  Thrombocytopenia: Phase II - Any Grade | 14.3
  Thrombocytopenia: Phase II - Grade 3/4 | 0
  Neutropenia: Phase I - Any Grade | 8.3
  Neutropenia: Phase I - Grade 3/4 | 0
  Neutropenia: Phase II - Any Grade | 4.8
  Neutropenia: Phase II - Grade 3/4 | 4.8
  Febrile Neutropenia: Phase I - Any Grade | 8.3
  Febrile Neutropenia: Phase I - Grade 3/4 | 8.3
  Febrile Neutropenia: Phase II - Any Grade | 0
  Febrile Neutropenia: Phase II - Grade 3/4 | 0
  Dizziness: Phase I - Any Grade | 8.3
  Dizziness: Phase I - Grade 3/4 | 8.3
  Dizziness: Phase II - Any Grade | 19
  Dizziness: Phase II - Grade 3/4 | 4.8
  Dyspnea: Phase I - Any Grade | 25
  Dyspnea: Phase I - Grade 3/4 | 8.3
  Dyspnea: Phase II - Any Grade | 33.3
  Dyspnea: Phase II - Grade 3/4 | 0
  Cough: Phase I - Any Grade | 25
  Cough: Phase I - Grade 3/4 | 0
  Cough: Phase II - Any Grade | 28.6
  Cough: Phase II - Grade 3/4 | 0
  Fatigue: Phase I - Any Grade | 33.3
  Fatigue: Phase I - Grade 3/4 | 0
  Fatigue: Phase II - Any Grade | 76
  Fatigue: Phase II - Grade 3/4 | 4.8
  Anorexia: Phase I - Any Grade | 33.3
  Anorexia: Phase I - Grade 3/4 | 0
  Anorexia: Phase II - Any Grade | 19
  Anorexia: Phase II - Grade 3/4 | 4.8
  Mucositis: Phase I - Any Grade | 41.7
  Mucositis: Phase I - Grade 3/4 | 0
  Mucositis: Phase II - Any Grade | 38
  Mucositis: Phase II - Grade 3/4 | 4.8
  Nausea: Phase I - Any Grade | 33.3
  Nausea: Phase I - Grade 3/4 | 0
  Nausea: Phase II - Any Grade | 28.6
  Nausea: Phase II - Grade 3/4 | 0
  Diarrhea: Phase I - Any Grade | 33.3
  Diarrhea: Phase I - Grade 3/4 | 0
  Diarrhea: Phase II - Any Grade | 33.3
  Diarrhea: Phase II - Grade 3/4 | 9.5
  Constipation: Phase I - Any Grade | 16.7
  Constipation: Phase I - Grade 3/4 | 0
  Constipation: Phase II - Any Grade | 23.8
  Constipation: Phase II - Grade 3/4 | 4.8
  Fever(no neutropenia): Phase I - Any Grade | 8.3
  Fever(no neutropenia): Phase I - Grade 3/4 | 0
  Fever(no neutropenia): Phase II - Any Grade | 19
  Fever(no neutropenia): Phase II - Grade 3/4 | 4.8
  Headache: Phase I - Any Grade | 50
  Headache: Phase I - Grade 3/4 | 0
  Headache: Phase II - Any Grade | 23.8
  Headache: Phase II - Grade 3/4 | 0
  Hypomagnesmia: Phase I - Any Grade | 0
  Hypomagnesmia: Phase I - Grade 3/4 | 0
  Hypomagnesmia: Phase II - Any Grade | 19
  Hypomagnesmia: Phase II - Grade 3/4 | 4.8
  Vomiting: Phase I - Any Grade | 16.7
  Vomiting: Phase I - Grade 3/4 | 0
  Vomiting: Phase II - Any Grade | 23.8
  Vomiting: Phase II - Grade 3/4 | 4.8

5. Secondary Outcome: Clinical Benefit Rate
Description: Clinical Benefit Rate (CR + PR + SD lasting more than 90 days)
Time Frame: 12 months
Population: Data was not collected or analyzed for this secondary objective.
Arm/Group | Pemetrexed + Cetuximab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Participants were monitored for adverse events for the duration of their participation in the trial, generally up to one year.
Description: Adverse Events are reported for all 36 participants that consented for the study, although 33 participants actually received treatment.
Arm/Group | Pemetrexed + Cetuximab
Serious Adverse Events (participants affected / at risk) | 11/36
Other Adverse Events (participants affected / at risk) | 32/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed + Cetuximab (N=36)
CNS CEREBROVASCULAR ISCHEMIA (Nervous system disorders) | 1 (1)
DEATH NOT ASSOCIATED WITH CTCAE TERM / DISEASE PROGRESSION NOS (General disorders) | 2 (2)
DEHYDRATION (Gastrointestinal disorders) | 1 (1)
DIZZINESS (Nervous system disorders) | 2 (2)
DYSPNEA (SHORTNESS OF BREATH) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
HEMORRHAGE, PULMONARY/UPPER RESPIRATORY / LUNG (Respiratory, thoracic and mediastinal disorders) | 1 (1)
INFECTION - OTHER (SPECIFY, __) (Infections and infestations) | 1 (1)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / BONE (OSTEOMYELITIS) (Infections and infestations) | 1 (1)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / LUNG (PNEUMONIA) (Infections and infestations) | 1 (1)
MAGNESIUM, SERUM-LOW (HYPOMAGNESEMIA) (Investigations) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 1 (1)
PNEUMONITIS/PULMONARY INFILTRATES (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PTT (PARTIAL THROMBOPLASTIN TIME) (Surgical and medical procedures) | 1 (1)
RASH: ACNE/ACNEIFORM (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed + Cetuximab (N=36)
ALBUMIN, SERUM-LOW (HYPOALBUMINEMIA) (Investigations) | 2 (2)
ALT, SGPT (SERUM GLUTAMIC PYRUVIC TRANSAMINASE) (Investigations) | 4 (9)
ANOREXIA (Gastrointestinal disorders) | 13 (18)
AST, SGOT(SERUM GLUTAMIC OXALOACETIC TRANSAMINASE) (Investigations) | 3 (12)
AUDITORY/EAR - OTHER (Ear and labyrinth disorders) | 1 (2)
BILIRUBIN (HYPERBILIRUBINEMIA) (Investigations) | 1 (2)
BRONCHOSPASM, WHEEZING (Respiratory, thoracic and mediastinal disorders) | 1 (1)
CALCIUM, SERUM-LOW (HYPOCALCEMIA) (Investigations) | 1 (4)
COAGULATION - OTHER (Blood and lymphatic system disorders) | 1 (1)
CONFUSION (Nervous system disorders) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 7 (11)
CONSTITUTIONAL SYMPTOMS - OTHER (General disorders) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 11 (16)
DEHYDRATION (Gastrointestinal disorders) | 2 (2)
DERMATOLOGY/SKIN - OTHER (Skin and subcutaneous tissue disorders) | 1 (2)
DIARRHEA (Gastrointestinal disorders) | 8 (9)
DIZZINESS (Nervous system disorders) | 3 (3)
DRY SKIN (Skin and subcutaneous tissue disorders) | 2 (2)
DYSPNEA (SHORTNESS OF BREATH) (Respiratory, thoracic and mediastinal disorders) | 12 (22)
EDEMA: HEAD AND NECK (Blood and lymphatic system disorders) | 2 (2)
EDEMA: LIMB (Blood and lymphatic system disorders) | 2 (5)
EYELID DYSFUNCTION (Eye disorders) | 2 (2)
FATIGUE (ASTHENIA, LETHARGY, MALAISE) (General disorders) | 21 (57)
FEBRILE NEUTROPENIA (ANC <1.0 X 10E9/L, FEVER >=38.5 DEGREES C) (Infections and infestations) | 1 (1)
FEVER (IN THE ABSENCE OF NEUTROPENIA, WHERE NEUTROPENIA IS DEFINED AS ANC <1.0 X 10E9/L) (General disorders) | 6 (9)
GASTROINTESTINAL - OTHER (Gastrointestinal disorders) | 3 (3)
GLUCOSE, SERUM-HIGH (HYPERGLYCEMIA) (Investigations) | 2 (2)
HAIR LOSS/ALOPECIA (SCALP OR BODY) (Skin and subcutaneous tissue disorders) | 8 (12)
HEARTBURN/DYSPEPSIA (Gastrointestinal disorders) | 6 (8)
HEMOGLOBIN (Blood and lymphatic system disorders) | 4 (8)
HEMOLYSIS (E.G., IMMUNE HEMOLYTIC ANEMIA, DRUG-RELATED HEMOLYSIS) (Blood and lymphatic system disorders) | 1 (1)
HEMORRHAGE, GI / ANUS (Gastrointestinal disorders) | 1 (1)
HEMORRHAGE, PULMONARY/UPPER RESPIRATORY / LUNG (Respiratory, thoracic and mediastinal disorders) | 1 (1)
HEMORRHAGE, PULMONARY/UPPER RESPIRATORY / NOSE (Respiratory, thoracic and mediastinal disorders) | 2 (2)
HEMORRHAGE/BLEEDING - OTHER (General disorders) | 1 (1)
HEMORRHOIDS (Gastrointestinal disorders) | 1 (1)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
INFECTION WITH GRADE 3 OR 4 NEUTROPHILS (ANC <1.0 X 10E9/L) / UNGUAL (NAILS) (Infections and infestations) | 1 (1)
INFECTION - OTHER (Infections and infestations) | 1 (1)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / CONJUNCTIVA (Infections and infestations) | 2 (2)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / MUCOSA (Infections and infestations) | 1 (1)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / SKIN (CELLULITIS) (Infections and infestations) | 2 (2)
INSOMNIA (General disorders) | 4 (6)
LEUKOCYTES (TOTAL WBC) (Blood and lymphatic system disorders) | 2 (2)
MAGNESIUM, SERUM-LOW (HYPOMAGNESEMIA) (Investigations) | 3 (3)
METABOLIC/LABORATORY - OTHER (Investigations) | 2 (7)
MOOD ALTERATION / AGITATION (Psychiatric disorders) | 1 (1)
MOOD ALTERATION / ANXIETY (Psychiatric disorders) | 3 (4)
MOOD ALTERATION / DEPRESSION (Psychiatric disorders) | 1 (2)
MUCOSITIS/STOMATITIS (CLINICAL EXAM) / ORAL CAVITY (Surgical and medical procedures) | 11 (17)
MUCOSITIS/STOMATITIS (CLINICAL EXAM) / PHARYNX (Surgical and medical procedures) | 1 (1)
MUSCLE WEAKNESS, GENERALIZED OR SPECIFIC AREA (NOT DUE TO NEUROPATHY) / EXTREMITY-LOWER (Musculoskeletal and connective tissue disorders) | 1 (3)
MUSCLE WEAKNESS, GENERALIZED OR SPECIFIC AREA (NOT DUE TO NEUROPATHY) / WHOLE BODY/GENERALIZED (Musculoskeletal and connective tissue disorders) | 1 (1)
NAIL CHANGES (Skin and subcutaneous tissue disorders) | 4 (6)
NAUSEA (Gastrointestinal disorders) | 10 (23)
NEUROPATHY: CRANIAL / CN VIII HEARING AND BALANCE (Nervous system disorders) | 1 (1)
NEUROPATHY: SENSORY (Nervous system disorders) | 8 (9)
NEUTROPHILS/GRANULOCYTES (ANC/AGC) (Blood and lymphatic system disorders) | 2 (3)
OBSTRUCTION/STENOSIS OF AIRWAY / BRONCHUS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTITIS, EXTERNAL EAR (NON-INFECTIOUS) (Ear and labyrinth disorders) | 1 (1)
PAIN / ABDOMEN NOS (Gastrointestinal disorders) | 3 (4)
PAIN / BACK (General disorders) | 1 (2)
PAIN / BONE (Musculoskeletal and connective tissue disorders) | 2 (4)
PAIN / CHEST WALL (Respiratory, thoracic and mediastinal disorders) | 1 (2)
PAIN / CHEST/THORAX NOS (Respiratory, thoracic and mediastinal disorders) | 3 (4)
PAIN / FACE (General disorders) | 1 (1)
PAIN / HEAD/HEADACHE (General disorders) | 9 (10)
PAIN / JOINT (Musculoskeletal and connective tissue disorders) | 2 (2)
PAIN / MUSCLE (Musculoskeletal and connective tissue disorders) | 1 (1)
PAIN / PLEURA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PAIN / TUMOR PAIN (General disorders) | 1 (2)
PAIN / URETHRA (Renal and urinary disorders) | 1 (1)
PAIN - OTHER (General disorders) | 2 (2)
PERICARDIAL EFFUSION (NON-MALIGNANT) (Cardiac disorders) | 1 (1)
PHLEBITIS (INCLUDING SUPERFICIAL THROMBOSIS) (Vascular disorders) | 1 (3)
PLATELETS (Blood and lymphatic system disorders) | 4 (7)
PNEUMONITIS/PULMONARY INFILTRATES (Respiratory, thoracic and mediastinal disorders) | 1 (1)
POTASSIUM, SERUM-LOW (HYPOKALEMIA) (Investigations) | 2 (2)
PROCTITIS (Gastrointestinal disorders) | 1 (1)
PRURITUS/ITCHING (Skin and subcutaneous tissue disorders) | 8 (10)
PULMONARY/UPPER RESPIRATORY - OTHER (Respiratory, thoracic and mediastinal disorders) | 1 (1)
RASH/DESQUAMATION (Skin and subcutaneous tissue disorders) | 3 (6)
RASH: ACNE/ACNEIFORM (Skin and subcutaneous tissue disorders) | 18 (56)
RASH: HAND-FOOT SKIN REACTION (Skin and subcutaneous tissue disorders) | 1 (3)
RIGORS/CHILLS (General disorders) | 1 (1)
SKIN BREAKDOWN/DECUBITUS ULCER (Skin and subcutaneous tissue disorders) | 2 (3)
SODIUM, SERUM-LOW (HYPONATREMIA) (Investigations) | 2 (2)
SUPRAVENTRICULAR AND NODAL ARRHYTHMIA / ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1)
SUPRAVENTRICULAR AND NODAL ARRHYTHMIA / ATRIAL TACHYCARDIA/PAROXYSMAL ATRIAL TACHYCARDIA (Cardiac disorders) | 1 (1)
SUPRAVENTRICULAR AND NODAL ARRHYTHMIA / SINUS TACHYCARDIA (Cardiac disorders) | 2 (2)
SWEATING (DIAPHORESIS) (General disorders) | 1 (1)
TASTE ALTERATION (DYSGEUSIA) (Gastrointestinal disorders) | 5 (8)
TREMOR (Nervous system disorders) | 1 (1)
URINARY FREQUENCY/URGENCY (Renal and urinary disorders) | 2 (2)
URTICARIA (HIVES, WELTS, WHEALS) (Skin and subcutaneous tissue disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 7 (8)
WEIGHT LOSS (General disorders) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No